CLINICAL TRIAL: NCT06954038
Title: A Randomized, Double Dummy, Placebo-controlled Pilot Study to Evaluate the Beneficial Effects of an Oral Nutritional Supplement Based on Leonurus Cardiaca for the Improvement of Mood and Anxiety
Brief Title: Evaluate the Beneficial Effects of an Oral Nutritional Supplement Based on Leonurus Cardiaca for the Improvement of Mood and Anxiety
Acronym: LEONORUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2312/01092024; Leonurus (Other: University of Pavia)
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: General Anxiety Disorder
Keywords: Leonurus cardiaca; Herbal extract; Anxiety; SCAG scale; Herbal remedy for GAD; HAM-A; PSQ; SF-12
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leonurus 250 mg (Experimental): Participants in this arm will receive a standardized oral supplement containing 250 mg of Leonurus cardiaca formulated in phospholipids, taken once daily in the morning for 30 days.
  Interventions: Dietary Supplement: Leonurus cardiaca extract 250 mg
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo identical in appearance to the active supplement, taken once daily in the morning for 30 days.
  Interventions: Dietary Supplement: Placebo
- Leonurus 500 mg (Experimental): Participants in this arm will receive a standardized oral supplement containing 500 mg of Leonurus cardiaca formulated in phospholipids, taken once daily in the morning for 30 days.
  Interventions: Dietary Supplement: Leonurus cardiaca extract 500 mg

INTERVENTIONS:
Dietary Supplement: Leonurus cardiaca extract 250 mg — Participants will receive a dietary supplement containing 250 mg of Leonurus cardiaca extract formulated in phospholipids. The supplement is administered as a single oral capsule, once daily in the morning, for 30 consecutive days.
  Arms: Leonurus 250 mg
Dietary Supplement: Placebo — Participants will receive a placebo capsule identical in appearance to the active supplement, administered twice daily for 30 consecutive days.
  Arms: Placebo
Dietary Supplement: Leonurus cardiaca extract 500 mg — Participants will receive a dietary supplement containing 500 mg of Leonurus cardiaca extract formulated in phospholipids. The supplement is administered as a single oral capsule, once daily in the morning, for 30 consecutive days.
  Arms: Leonurus 500 mg

SUMMARY:
This study aims to evaluate the efficacy and safety of Leonurus cardiaca extract in reducing anxiety symptoms in adults with Generalized Anxiety Disorder (GAD). Sixty drug-free participants aged 20-50 years with a diagnosis of GAD will be randomly assigned to receive either Leonurus cardiaca extract or placebo for 30 days. The primary outcome is the reduction in anxiety symptoms assessed by the SCAG scale. Secondary outcomes include changes in quality of life (SF-12), perceived stress (PSQ), anxiety severity (HAM-A), and anthropometric measures. Safety will be assessed through liver, kidney, and thyroid function tests. Assessments will be conducted at baseline, day 14, and day 30.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 50 years
* Diagnosis of a generalised anxiety disorder (GAD), with manifestations occurring for >= 6 months that include excessive worry, poor concentration, restlessness, muscle tension, irritability, fatigue and difficulty sleeping

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Use of hormonal contraceptives in the last 3 months
* Current diagnosis of major psychiatric disorders (e.g., major depressive disorder, severe anxiety disorders, schizophrenia, bipolar disorder)
* Known endocrine disorders (e.g., hypothyroidism, hyperthyroidism, diabetes)
* Use of medications that could affect mood or the menstrual cycle (e.g., SSRIs, anxiolytics, antipsychotics)
* Severe hepatic or renal impairment
* Any other serious or unstable medical condition that, in the investigator's judgment, could interfere with study participation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in SCAG (Sandoz Clinical Assessment-Geriatric) score | Baseline, week 1 and week 4
  Anxiety and neurovegetative symptoms will be assessed using the SCAG scale at baseline, 14 days, and 30 days. The SCAG includes items scored from 0 (absent) to 4 (very severe), providing a composite measure of mood, anxiety, headache, and sleep quality.

SECONDARY OUTCOMES:
Change in Perceived Stress Questionnaire (PSQ) score | Baseline, week 1 and week 4
  Stress perception will be assessed across four domains (worries, tension, joy, and demands) using the PSQ ( Perceived Stress Questionnaire), a 14-item survey. The total score ranges from a minimum of 0 to a maximum of 56. Higher scores on the scale indicate higher perceived stress and generally reflect a worse outcome in terms of stress-related well-being.
Change in Hamilton Anxiety Rating Scale (HAM-A) score | Baseline, week 1 and week 4
  The severity of anxiety symptoms will be evaluated using the HAM-A scale, which consists of 14 items each scored from 0 to 4. Total score ranges from 0 (no anxiety) to 56 (severe anxiety).
Change in SF-12 Health Survey score | Baseline, week 1 and week 4
  The Short Form Health Survey (SF-12) will be used to evaluate physical and mental well-being. Two summary scores (Physical and Mental Component) will be analyzed. It measures health status through summary scores for the physical (PCS-12) and mental (MCS-12) components. PCS-12 and MCS-12 summary scores are standardised to have mean 50 and standard deviation 10 in the general US population
Change in body weight | Baseline and week 4
  Body weight (kg) will be measured at baseline and at day 30.
Change in Body Mass Index (BMI) | Baseline and week 4
  BMI (kg/m²) will be calculated from measured weight and height at baseline and after 30 days.
Change in liver function tests (AST, ALT, gamma-GT) | Baseline and week 4
  Blood tests will be performed at baseline and after 30 days to monitor liver safety through AST, ALT, and GGT levels (U/L).
Change in creatinine levels | Baseline and week 4
  Serum creatinine will be measured at baseline and day 30 to assess renal function.
Change in thyroid-stimulating hormone (TSH) levels | Baseline and week 4
  Thyroid-stimulating hormone (TSH) levels will be evaluated through blood samples collected at baseline and after 30 days to assess the effect of the intervention on pituitary-thyroid axis activity.
Change in free triiodothyronine (FT3) levels | Baseline and week 4
  Free triiodothyronine (FT3) levels will be assessed through blood samples collected at baseline and after 30 days to evaluate peripheral thyroid hormone activity.
Change in free thyroxine (FT4) levels | Baseline and week 4
  Free thyroxine (FT4) levels will be assessed from blood samples taken at baseline and after 30 days in order to monitor thyroid gland function.
Change in Cortisol levels | Baseline, week 1 and week 4
  Salivary cortisol assessment: 3 evaluation tests on the day x 3 times (first visit = baseline, after 7 days, after 28 days)

IPD SHARING:
Plan to Share IPD: No